CLINICAL TRIAL: NCT05124730
Title: Open, Comparative, Randomized, Crossover, Single Dose Bioequivalence Study of Metformin 500 mg Prolonged Release Tablets (JSC Farmak, Ukraine) vs Glucophage® XR 500 mg Prolonged Release Tablets in Healthy Subjects Under Fasting Conditions.
Brief Title: Fasting Bioequivalence Study of 2 Metformin 500 mg Prolonged Release Tablets in 44 Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joint Stock Company "Farmak" (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FK/MTF/500/2021
Record Dates: First submitted 2021-11-09; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Pharmacokinetics
Keywords: bioequivalence; pharmacokinetics; generic drugs; Metformin 500 mg Prolonged Release Tablets; Prolonged Release Tablets; oral dosage form
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Masking Description: The study was open-labelled; however, analysts did not have access to the randomization scheme to prevent bias during analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Metformin 500 mg Prolonged Release Tablets (JSC Farmak, Ukraine)
  Interventions: Drug: Metformin 500mg prolonged release tablets (JSC Farmak, Ukraine)
- Treatment B (Active Comparator): Glucophage® XR 500 mg prolonged release tablets (Merck Serono Ltd, UK)
  Interventions: Drug: Glucophage® XR 500 mg prolonged release tablets (Merck Serono Ltd, UK)

INTERVENTIONS:
Drug: Metformin 500mg prolonged release tablets (JSC Farmak, Ukraine) — One tablet of the Test product was administered orally with 240 mL of water.
  Other Names: Diaformin® SR (sustained-release) 500mg tablets (JSC Farmak, Ukraine); Diabufor® XR 500mg tablets (JSC Farmak, Ukraine)
  Arms: Treatment A
Drug: Glucophage® XR 500 mg prolonged release tablets (Merck Serono Ltd, UK) — One tablet of Reference (R) Product was administered orally with 240 mL of water.
  Arms: Treatment B

SUMMARY:
This study was designed to compare the bioavailability of the Test Product Metformin 500mg Prolonged Release Tablets (JSC Farmak, Ukraine) and Reference Product Glucophage® XR 500 mg Prolonged Release Tablets (Merck Serono Ltd, UK) in healthy male and female volunteers under fasting conditions.

DETAILED DESCRIPTION:
An Open, Comparative, Randomized, Crossover Clinical Trial to Evaluate the Bioequivalence of Single Doses of Test Product Metformin 500mg Prolonged Release Tablets (JSC Farmak, Ukraine) and Reference Product Glucophage® XR 500 mg Prolonged Release Tablets (Merck Serono Ltd, UK) in Healthy, Adult Male and Female Subjects under Fasting Conditions.

During each period 21 blood samples were taken: prior to dosing (-1.0) and 1.0, 2.0, 3.0, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 8.5, 9.0, 10.0, 12.0, 16.0, 24.0, 32.0 and 36.0 hours after Investigational Medicinal Product (IMP) administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and non-pregnant and no breast-feeding females (must have a negative pregnansy test result prior to dosing). Caucasian race.
* Non-smoker or past-smoker (who has stopped smoking at least 6 months before the first dosing).
* Body Mass Index (BMI) 18.5 to 30.0 kg/m2, inclusive and body weight between 50 kg and 100 kg (on the day of screening).
* Subject was available for the whole study and has provided his/her written informed consent.
* Subjects in good health, as determined by screening medical history, physical examination, vital signs assessments (pulse rate, systolic and diastolic blood pressure, and body temperature) and 12-lead ECG. Minor deviations outside the reference ranges were acceptable, if deemed not clinically significant by the Investigator.
* All laboratory screening results within the normal range. Minor deviations outside the reference ranges were acceptable, if deemed not clinically significant by the Clinical Investigator.
* Acceptance of use of contraceptive measures during the whole study by both female and male subjects.

Exclusion Criteria:

* Known cardiovascular disease, history of hypotension.
* Factors in the subject's history that may predispose to ketoacidosis (including pancreatic insulin deficiency, history of pancreatitis, caloric restriction disorders, restricted food intake, alcohol abuse).
* Gastrointestinal, renal or hepatic diseases and/or pathological findings present or in history, which might interfere with the drug pharmacokinetics.
* Glucose level out of the limit 3.3 mmol/L - 5.5 mmol/Lat screening, as determined by screening clinical laboratory evaluations.
* Previous liver disease or clinically significant elevations in serum transaminases at the screening.
* Acute or chronic diseases and/or clinical finding which may interfere with the aims of the study or with the drug's safety, tolerability, bioavailability and/or pharmacokinetics of the IMP.
* History of kidney disease and with impaired renal function.
* History of severe allergy or allergic reactions to the study IMP, its excipients or related drugs.
* Clinically significant illness within 28 days before the first dosing, including major surgery.
* Any significant clinical abnormality including Hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), and / or (human immunodeficiency virus) HIV. (On screening).
* Positive result of blood pregnancy test at screening or positive urine pregnancy test at check-in or breast-feeding or lack of results of pregnancy test.
* Positive results of drugs of abuse in urine at screening and at check-in.
* Positive result of alcohol breath test at screening and at check-in.
* Positive result of urine cotinine test at screening and at check-in.
* Serious mental disease and/or inability to cooperate with clinical team.
* Sitting blood pressure after a minimum of 5 minutes of rest is out of the range of 90-140 mmHg for systolic blood pressure (BP) and/or 60-90 mmHg for diastolic BP and/or heart rate out of the range of 50-100 bpm during the screening procedure.
* Body ear temperature is out of the range of 35.7 - 37.3°C at screening and at check-in.
* Orthostatic hypotension during the screening procedure.
* Drug, alcohol (of ≥ 40 g per day pure ethanol), solvents or caffeine abuse.
* Use of organ-toxic drugs or systemic drugs known to substantially alter liver metabolism within 90 days before the first dosing.
* Use of any prescription medication for a period of 28 days before the first dosing.
* Use of any OTC (over-the-counter) medication including vitamins, herbal medications and food supplements less than 14 days before the first dosing.
* Getting a tattoo, body piercing or any cosmetic treatment involving skin piercing within 90 days before the screening unless evaluated by Investigator as non-significant for inclusion in the study.
* Donation or loss of at least 500 mL of blood within 90 days or donation of plasma or platelets within 14 days before the first dosing.
* Anemia, haemoglobin below 120 g/L for women and 130 g/L for men at screening.
* Less than 30 days between exit procedure in previous study and the first dosing in in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2021-05-29 (Actual); Study Completion 2021-05-29 (Actual)

PRIMARY OUTCOMES:
AUC0-t | up to 36 hours post-administration
  Area under the plasma drug concentration versus time curve
Cmax | up to 36 hours post-administration
  Maximum plasma concentration observed.

SECONDARY OUTCOMES:
AUC(0-∞) | up to 36 hours post-administration
  Area under the plasma drug concentration versus time curve from time zero to infinity
AUC(0-12h) | from time zero to time 12 hours after dosing.
  The area under the plasma drug concentration versus time curve calculated from time zero to time 12 hours after dosing.
AUC(12h-t) | from time 12 hours after dosing up to 36 hours post-administration
  The area under the plasma drug concentration versus time curve calculated from time 12 hours after dosing to time of the last sample above LLOQ
AUC(0-24h) | from time zero to time 24 hours after dosing
  The area under the plasma drug concentration versus time curve calculated from time zero to time 24 hours after dosing.
tmax | up to 36 hours post-administration
  the time of the maximum plasma drug concentration.
λz | up to 36 hours post-administration
  Apparent first-order elimination
t1/2 | up to 36 hours post-administration
  The elimination or terminal half-life
AUCres | up to 36 hours post-administration
  Residual area

CONTACTS AND LOCATIONS:
Overall Officials: Vlad Udovytskyi, Study Chair — Joint Stock Company "Farmak"
Locations (1):
- QUINTA-ANALYTICA s.r.o., Prague, Czechia

IPD SHARING:
Plan to Share IPD: No